CLINICAL TRIAL: NCT01176344
Title: Does Vitamin D Supplementation Prevent Progression of Knee Osteoarthritis? A Randomised Controlled Trial
Brief Title: VItamin D Effect on Osteoarthritis Study
Acronym: VIDEO
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Menzies Institute for Medical Research (Other)
Collaborators: Monash University (Other)
Responsible Party: Principal Investigator, Changhai Ding, Professor, Menzies Institute for Medical Research
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VIDEO605501
Record Dates: First submitted 2010-08-04; First posted 2010-08-06 (Estimated); Last update posted 2015-09-09 (Estimated); Status verified 2015-09

CONDITIONS: Osteoarthritis, Knee
Keywords: Vitamin D supplementation; Osteoarthritis; Knee; Randomised clinical trial (RCT); Cartilage; MRI
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis | interventions — Vitamin D

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vitamin D supplementation (Experimental): Participants in the intervention arm will receive 50,000 IU (1.25 mg) cholecalciferol capsules given once monthly
  Interventions: Drug: Vitamin D
- Placebo (Placebo Comparator): The control arm will receive identical inert placebo capsules given once monthly.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Vitamin D — 50,000 IU (1.25 mg) cholecalciferol capsules once monthly for 2 years
  Arms: Vitamin D supplementation
Drug: Placebo — Inert placebo capsules once monthly for 2 years.
  Arms: Placebo

SUMMARY:
Observational evidence suggests that vitamin D deficiency may have a role in the causes of osteoarthritis (OA) and there are biologically plausible mechanisms to explain this. There is, however, no evidence which shows that intervening with vitamin D supplementation can slow the progression of OA. This study is to determine if vitamin D supplementation can reduce knee pain and slow knee cartilage loss in OA patients comparing with a placebo. Use of MRI will provide sensitive measures of knee OA changes.

DETAILED DESCRIPTION:
Osteoarthritis (OA) is the most common joint disorder in the world. In 2004, OA was estimated to affect over 1.6 million Australians, with total costs of $1.4 billion. OA is the most frequent reason for joint replacement, at a cost of about $1 billion each year. Conventional treatment is palliative and costly, and currently there are no effective medical remedies for OA. These facts have led to 2000-2010 being labelled the Bone and Joint decade, and musculoskeletal disorders being recognised as a National Health Priority. The primary task for OA management should be to identify modifiable risk factors.

Vitamin D deficiency is very common in older people and has been linked with osteoporosis and falls in both older women and men. Emerging data suggests that it also plays an important role in the pathogenesis of knee OA. Firstly, vitamin D may have direct effects on chondrocytes in osteoarthritic cartilage; secondly, chronic vitamin D inadequacy in adults has adverse effects on calcium metabolism, osteoblast activity, matrix ossification and bone density, and thus could impair the ability of bone to respond optimally to pathophysiological processes in OA; and thirdly, low vitamin D levels are associated with loss of muscle strength and muscle mass in older men and women, which may be associated with an increased risk of knee OA. Some observational studies have shown that vitamin D insufficiency is associated with the progression and development of radiographic knee or hip OA. Recently we have demonstrated that baseline serum levels of 25-hydroxy-vitamin D(25-(OH)D) predicts change in cartilage volume in older adults over 2 years, and increases in vitamin D levels are associated with a further protective association. This suggests that vitamin D supplementation may enhance cartilage and bone health, and thus prevent disease progression in patients with knee OA.

The aim of this study is to compare the effects of vitamin D supplementation versus placebo on knee pain and knee structural changes in patients with symptomatic knee osteoarthritis over a 2- year period.

The proposed study design is a randomised, placebo-controlled, double-blind clinical trial. We will recruit 400 subjects (50-79 years old, having relatively good health and serum vitamin D level of <60 and >12.5 nmol/L) with symptomatic knee OA for at least 6 months using a combined strategy in Southern Tasmania and Melbourne. Participants in the intervention arm (n=200) will receive 50,000 IU (1.25 mg) cholecalciferol tablets given once monthly, whilst those in the control arm (n=200) will receive an identical inert placebo. All participants will be provided recommended standard of care. Knee structural changes including knee cartilage volume, cartilage defects, tibial bone area, bone marrow lesions, and meniscal pathology (assessed by MRI), and knee pain at baseline and 2 years later will be determined as outcome measures. Other explanatory factors, such as serum vitamin D levels, height, weight, physical activity, and smoking will also be determined through study period.

Significance:

Observational evidence suggests that vitamin D deficiency may have a role in the progression of OA and there are biologically plausible mechanisms to explain this. However, randomized controlled trials using a sensitive method are required to determine whether intervening with vitamin D supplementation can in fact slow the progression of this disease. In this study, the randomized, placebo-controlled, double-blind design, and the use of MRI to provide sensitive and precise measures of knee structural change will ensure a rigorous evaluation of the impact of vitamin D supplementation on knee OA. It will be the first long term clinical trial to determine comprehensively the effects on knee structural changes (cartilage, bone) utilizing the pioneering MRI techniques and limb muscle strength assessment. This study builds upon previous clinical and epidemiological studies that supports the objectives of the Bone and Joint Decade organization and addresses a National Health Priority Area.

ELIGIBILITY:
Inclusion Criteria:

1. Age 50-79 years old;
2. Men and women with symptomatic knee osteoarthritis (OA) with a pain visual analogue scale (VAS) of at least 20 mm in most days of the last month;
3. Have an American College of Rheumatology (ACR) functional class rating of I, II and III;
4. Have relatively good health (0-2 according to the investigator's global assessment of disease status on a 5-point Likert scale, range 0 [very well] to 4 [very poor]);
5. Have serum vitamin D level of >12.5 nmol/L and <60 nmol/L;
6. Are able to read, speak and understand English, capable of understanding the study requirements and willing to co-operate with the study instructions;
7. Are able and willing to give informed consent;
8. Are willing and able to give blood samples;
9. Are willing and able to have knee MRIs performed

Exclusion Criteria:

1. Have Grade 3 radiographic changes in their knee which is to be investigated;
2. Have severe knee pain (more than 80 mm on a 100-mm visual analogue scale,VAS) in most days of the last month;
3. Have any contra-indications for having MRIs scans performed;
4. Have had significant trauma to the knees including arthroscopy or significant injury to ligaments or menisci of the knee within 1 year preceding the screening visit;
5. Have ever had knee joint replacement;
6. Have anticipated need for knee or hip surgery in the next 2 years;
7. Have any stomach or intestinal condition possibly affecting oral drug absorption;
8. Have any clinically significant condition(s) such as (but not limited to) rheumatoid arthritis, psoriatic arthritis, lupus, active cancer, cardiac or renal function impairment or hypersensitivity to vitamin D that in the opinion of the investigator may compromise their safety or compliance, interfere with evaluation or preclude completion of the study.

Ages: 50 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 413 (Actual)
Dates: Start 2010-08; Primary Completion 2013-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Loss of knee cartilage volume | Over 2 years (Cartilage volume will be assessed at baseline and 2 years later)
  Cartilage volume will be assessed using magnetic resonance imaging (MRI)
Change in knee pain | Over 2 years
  Assessed using WOMAC

SECONDARY OUTCOMES:
Progression of knee cartilage defects | Over 2 years (Cartilahe defects will be measured at baseline and 2 years later)
  Knee cartilage defects will be measured using MRI.
Change in bone marrow lesions | Over 2 years
  Assessed using MRI
Change in knee pain | Over 2 years
  Assessed using VAS
Change in physical function | Over 2 years
  Assessed using WOMAC function
Change in joint effusion | Over 2 years
  Assessed using MRI
Central blood pressure | one year
  Radial applanation tonometry
Aortic stiffness | one year
  Carotid to femoral pulse wave velocity

CONTACTS AND LOCATIONS:
Overall Officials: Changhai Ding, MD, Principal Investigator — Menzies Research Institute & Monash University; Graeme Jones, MD, Principal Investigator — Menzies Institute for Medical Research; Flavia M Cicuttini, PhD, Principal Investigator — Monash University
Locations (2):
- Australia (2):
  - Menzies Research Institute, University of Tasmania, Hobart, Tasmania
  - Department of Epidemiology & Preventive Medicine, Monash University, Melbourne, Victoria

REFERENCES:
- [Background] Ding C, Cicuttini F, Parameswaran V, Burgess J, Quinn S, Jones G. Serum levels of vitamin D, sunlight exposure, and knee cartilage loss in older adults: the Tasmanian older adult cohort study. Arthritis Rheum. 2009 May;60(5):1381-9. doi: 10.1002/art.24486. PMID 19404958
- [Derived] Wang T, Zheng S, Jin X, Cen H, Zhu Z, Han W, Wluka A, Cicuttini F, Cao P, Ding C. Baseline 25-hydroxyvitamin D levels predict the effects of vitamin D supplementation on joint symptoms and cartilage loss in patients with knee osteoarthritis. Rheumatol Adv Pract. 2025 May 27;9(3):rkaf061. doi: 10.1093/rap/rkaf061. eCollection 2025. PMID 40677617
- [Derived] Chang J, Chen T, Yan Y, Zhu Z, Han W, Zhao Y, Antony B, Wluka A, Winzenberg T, Cicuttini F, Ding C. Associations between the morphological parameters of proximal tibiofibular joint (PTFJ) and changes in tibiofemoral joint structures in patients with knee osteoarthritis. Arthritis Res Ther. 2022 Jan 27;24(1):34. doi: 10.1186/s13075-022-02719-8. PMID 35086561
- [Derived] Zheng S, Tu L, Cicuttini F, Zhu Z, Han W, Antony B, Wluka AE, Winzenberg T, Aitken D, Blizzard L, Jones G, Ding C. Depression in patients with knee osteoarthritis: risk factors and associations with joint symptoms. BMC Musculoskelet Disord. 2021 Jan 7;22(1):40. doi: 10.1186/s12891-020-03875-1. PMID 33413273
- [Derived] Tu L, Zheng S, Cicuttini F, Jin X, Han W, Zhu Z, Antony B, Winzenberg T, Jones G, Gu J, Wluka AE, Ding C. Effects of Vitamin D Supplementation on Disabling Foot Pain in Patients With Symptomatic Knee Osteoarthritis. Arthritis Care Res (Hoboken). 2021 Jun;73(6):781-787. doi: 10.1002/acr.24371. PMID 32623812
- [Derived] Cuellar WA, Blizzard L, Hides JA, Callisaya ML, Jones G, Cicuttini F, Wluka AE, Ding C, Winzenberg TM. Vitamin D supplements for trunk muscle morphology in older adults: secondary analysis of a randomized controlled trial. J Cachexia Sarcopenia Muscle. 2019 Feb;10(1):177-187. doi: 10.1002/jcsm.12364. Epub 2018 Nov 22. PMID 30565892
- [Derived] Wang X, Jin X, Blizzard L, Antony B, Han W, Zhu Z, Cicuttini F, Wluka AE, Winzenberg T, Jones G, Ding C. Associations Between Knee Effusion-synovitis and Joint Structural Changes in Patients with Knee Osteoarthritis. J Rheumatol. 2017 Nov;44(11):1644-1651. doi: 10.3899/jrheum.161596. Epub 2017 Sep 1. PMID 28864651
- [Derived] Zhu Z, Otahal P, Wang B, Jin X, Laslett LL, Wluka AE, Antony B, Han W, Wang X, Winzenberg T, Cicuttini F, Jones G, Ding C. Cross-sectional and longitudinal associations between serum inflammatory cytokines and knee bone marrow lesions in patients with knee osteoarthritis. Osteoarthritis Cartilage. 2017 Apr;25(4):499-505. doi: 10.1016/j.joca.2016.10.024. Epub 2016 Nov 9. PMID 27836676
- [Derived] Jin X, Jones G, Cicuttini F, Wluka A, Zhu Z, Han W, Antony B, Wang X, Winzenberg T, Blizzard L, Ding C. Effect of Vitamin D Supplementation on Tibial Cartilage Volume and Knee Pain Among Patients With Symptomatic Knee Osteoarthritis: A Randomized Clinical Trial. JAMA. 2016 Mar 8;315(10):1005-13. doi: 10.1001/jama.2016.1961. PMID 26954409
- [Derived] Zhu Z, Jin X, Wang B, Wluka A, Antony B, Laslett LL, Winzenberg T, Cicuttini F, Jones G, Ding C. Cross-Sectional and Longitudinal Associations Between Serum Levels of High-Sensitivity C-Reactive Protein, Knee Bone Marrow Lesions, and Knee Pain in Patients With Knee Osteoarthritis. Arthritis Care Res (Hoboken). 2016 Oct;68(10):1471-7. doi: 10.1002/acr.22834. Epub 2016 Sep 6. PMID 26748954
- [Derived] Veloudi P, Blizzard CL, Ding CH, Cicuttini FM, Jin X, Wluka AE, Winzenberg T, Jones G, Sharman JE. Effect of Vitamin D Supplementation on Aortic Stiffness and Arterial Hemodynamics in People With Osteoarthritis and Vitamin D Deficiency. J Am Coll Cardiol. 2015 Dec 15;66(23):2679-2681. doi: 10.1016/j.jacc.2015.10.007. No abstract available. PMID 26670070
- [Derived] Cao Y, Jones G, Cicuttini F, Winzenberg T, Wluka A, Sharman J, Nguo K, Ding C. Vitamin D supplementation in the management of knee osteoarthritis: study protocol for a randomized controlled trial. Trials. 2012 Aug 6;13:131. doi: 10.1186/1745-6215-13-131. PMID 22867111